CLINICAL TRIAL: NCT02163538
Title: A Comparison of Industry Leading Energy Devices for Use in Gynecologic Laparoscopy: Articulating Enseal Versus Ligasure Energy Devices
Brief Title: Articulating Enseal Versus Ligasure Energy Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Resad Pasic, Professor with Tenure of Obstetrics and Gynecology, University of Louisville
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Energy Devices-UL
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2018-01-17 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-11

CONDITIONS: Task Performance
Keywords: energy device; laparoscopic; hysterectomy; enseal; ligasure; raw tlx

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- articulating Enseal (Active Comparator): This group of women undergoing total laparoscopic hysterectomy is randomized to the the articulating Enseal energy device.
  Interventions: Device: articulating Enseal
- Ligasure device (Active Comparator): This group of women undergoing hysterectomy is randomized to the Ligasure energy device.
  Interventions: Device: Ligasure device

INTERVENTIONS:
Device: articulating Enseal — Vessel-sealing device used for laparoscopic hysterectomy.
  Arms: articulating Enseal
Device: Ligasure device — Vessel-sealing device used for laparoscopic hysterectomy.
  Arms: Ligasure device

SUMMARY:
This is an exploratory study to assess the ability of the raw-TLX (raw Task Load Index) ergonomic assessment tool to detect differences in surgeon workload when using commercially available advanced bipolar devices. It is anticipated that the raw-TLX version of the validated NASA-TLX ergonomic assessment tool will detect less surgeon effort required in the procedure when articulating ENSEAL is utilized. The Articulating ENSEAL device may also positively impact other variables such as blood loss, operative time and cost.

DETAILED DESCRIPTION:
This study is a single-center, single-blinded, randomized control, pilot trial that will be conducted at the University of Louisville Hospital. It is designed to assess whether there are different surgical outcomes with regard to surgeon perception of ease of instrument use, operative time, estimated blood loss, cost and perioperative complication rates between the Ethicon Articulating Enseal versus the LigaSure for total laparoscopic hysterectomy. This will be assessed using the raw-TLX version of the validated NASA-TLX scale.

The study will be single-blinded in that the patient will not be informed of their group assignment; it is impossible to blind the surgeon using the devices.

Methods and Procedures:

Patients undergoing total laparoscopic hysterectomy will be recruited from our University of Louisville Health Care Outpatient Center (HCOC) outpatient office and will be consented for participation in the study during their preoperative office visit.

Patients will be randomized pre-operatively on their date of surgery to one of two groups:

Group 1: The articulating Enseal device will be used during the hysterectomy. Group 2: The Ligasure device will be used during the hysterectomy.

All cases will be videotaped for review of operative time and complications; this is standard procedure at our institution.

To evaluate our primary objective, i.e., the potential ergonomic and surgical advantages of an articulating tip in an energy device, the raw-TLX of the validated NASA-TLX scale will be completed by the primary surgeon at the end of each surgery.

Subjects will be seen for study follow-up during their routine post-operative visits at 2 weeks, 6 weeks and within 3 months after surgery in the event of a hospital admission for a surgery-related complication.

No compensation for participation will be offered to patients and no compensation for subject recruitment will be gained by investigators. This will be disclosed during the informed consent process.

Inclusion Criteria:

* Age 18 or older
* Able and willing to provide informed consent
* Undergoing total laparoscopic hysterectomy

Exclusion Criteria:

* Under 18 years of age
* Severe endometriosis or adhesions requiring >15min of adhesiolysis prior to beginning hysterectomy
* Unsafe to use energy device due to decreased visualization or any other reason deemed to be unsafe by the surgeon
* Intra-operative decision to convert to laparotomy prior to use of energy device
* Current diagnosis of uterine, tubal ovarian or cervical malignancy.
* Patients who cannot read/understand English.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able and willing to provide informed consent
* Undergoing total laparoscopic hysterectomy

Exclusion Criteria:

* Under 18 years of age
* Severe endometriosis or adhesions requiring >15min of adhesiolysis prior to beginning hysterectomy
* Unsafe to use energy device due to decreased visualization or any other reason deemed to be unsafe by the surgeon intra-operative decision to convert to laparotomy prior to use of energy device
* Current diagnosis of uterine, tubal ovarian or cervical malignancy.
* Patients who cannot read/understand English.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Resad Pasic, MD, PhD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - University of Louisville Health Care Outpatient Center, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
Data shared with study sponsor, Ethicon, and will be submitted for journal publication.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Articulating Enseal | Ligasure Device
Started | 71 | 71
Completed | 70 | 70
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Articulating Enseal | Ligasure Device | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (6.9) | 41.3 (7.7) | 41.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Raw Task Load Index (TLX) Score Assigned by Surgeons
Description: The Official NASA Task Load Index (TLX) is a subjective workload assessment tool to allow users to perform subjective workload assessments on operator(s) working with various human-machine interface systems. By incorporating a multi-dimensional rating procedure, NASA TLX derives an overall workload score based on a weighted average of ratings on six subscales given below. The overall workload score ranges between 0 and 100 with 100 being the most demanding.
  Mental Demand Physical Demand Temporal Demand Performance Effort Frustration
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
units on a scale | 51.7 [39.6 to 59.0] | 32.5 [17.7 to 48.1]
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Intra- and Post-operative Complications
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
Participants | 1 | 2
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = 1.00, Chi-squared

3. Secondary Outcome: Estimated Blood Loss
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
mL | 100 [50 to 200] | 100 [50 to 150]
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = 0.582, Chi-squared

4. Secondary Outcome: Need for Second Energy Device Intra-operatively
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
Participants | 10 | 0
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = 0.0031, Chi-squared

5. Secondary Outcome: Time From Port Placement to Bilateral Uterine Artery Ligation and Hemostatsis.
Time Frame: During procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
minutes | 35 [25 to 48] | 30 [22 to 41]
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = 0.0281, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Time Required to Complete Procedure
Time Frame: End of surgery up to 4 hours
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Articulating Enseal | Ligasure Device
Number analyzed (Participants) | 70 | 70
Minutes | 97 [80 to 129] | 85 [69 to 120]
Statistical Analysis 1: Comparison: Articulating Enseal vs Ligasure Device; Test type: Superiority; p = .0821, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Articulating Enseal | Ligasure Device
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 2/70 | 1/70
Other Adverse Events (participants affected / at risk) | 0/70 | 0/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Articulating Enseal (N=70) | Ligasure Device (N=70)
blood transfusion (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
rectal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes